CLINICAL TRIAL: NCT04541628
Title: A Phase 1/2 Open-Label, Dose-Escalation, Safety, Tolerability, and Efficacy Study of SIG-001 in Adult Patients With Severe or Moderately-Severe Haemophilia A Without Inhibitors (SIG-001-121)
Brief Title: Safety & Efficacy of Encapsulated Allogeneic FVIII Cell Therapy in Haemophilia A
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: SIG-001 programme terminated
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Sigilon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIG-001-121
Record Dates: First submitted 2020-08-21; First posted 2020-09-09 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Hemophilia A
Keywords: Haemophilia A; Cell therapy; Gene therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SIG-001 (Experimental): Participants received a single dose of 50 milliliter (mL), 78.5 mL and 133 mL of SIG-001 spheres [an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce B-Domain Deleted Human Factor VIII (BDD-hFVIII) producing Spheres] administered laparoscopically into the peritoneal cavity.
  Interventions: Combination Product: SIG-001

INTERVENTIONS:
Combination Product: SIG-001 — Laparoscopic administration of SIG-001 spheres, an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce BDD-hFVIII.

SUMMARY:
SIG-001-121 is a first-in-human (FIH), phase 1/2, multi-centre, open-label, dose escalation study to assess the safety, tolerability, and preliminary efficacy of SIG-001 in adults with severe or moderately severe haemophilia A without inhibitors. Up to three dose cohorts (3 patients each) are planned. Cohort expansions (up to 3 additional patients) may be triggered to collect additional information about safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years or older
* Diagnosis of Haemophilia A defined as ≤2% FVIII activity
* Greater than 150 exposure days to treatment with FVIII products
* Use of reliable barrier contraception if applicable
* Normal levels of von Willebrand factor (VWF) antigen
* Able and willing to provide informed consent
* Willing to withdraw from FVIII prophylaxis during specified periods in the study

Exclusion Criteria:

* Body mass index (BMI) ≥35
* Current FVIII inhibitors (>0.6 Nijmegen Bethesda Units/mL) or prior Immune Tolerance Induction (ITI)
* History of allergic reaction or anaphylaxis to recombinant FVIII products or SIG-001 components
* Evidence of any bleeding disorder in addition to haemophilia A
* Abnormal laboratory values as defined in the protocol
* Active infection with Hepatitis B or Hepatitis C virus or currently managed with antiviral medications for Hepatitis B or C
* Uncontrolled HIV infection
* Active alcoholism or drug addiction during the 12 months before the screening visit
* Active malignancy or history of malignancy in the 5 years prior to study entry
* Participation in another investigational medicine or device study
* Prior administration of a gene therapy product
* Significant underlying disease or comorbidities that are a contraindication for general anaesthesia or laparoscopic procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Clinical Study Site, Indianapolis, Indiana
  - Clinical Study Site, Boston, Massachusetts
  - Clinical Study Site, Seattle, Washington
- United Kingdom (3):
  - Clinical Study Site, London
  - Clinical Study Site, Manchester
  - Clinical Study Site, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants received a single dose of 50 milliliter (mL) SIG-001 spheres [an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce B-Domain Deleted Human Factor VIII (BDD-hFVIII) producing Spheres] administered laparoscopically into the peritoneal cavity.
- Cohort 2: Participants received a single dose of 78.5 mL SIG-001 spheres [an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce BDD-hFVIII producing Spheres] administered laparoscopically into the peritoneal cavity.
- Cohort 3: Participants received a single dose of 133 mL SIG-001 spheres [an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce BDD-hFVIII producing Spheres] administered laparoscopically into the peritoneal cavity.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 1 | 1 | 1
Received at Least One Dose of Study Drug | 1 | 1 | 1
Completed | 0 | 0 | 0
Not Completed | 1 | 1 | 1
Not completed — Study Terminated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Cohort 1: Participants received a single dose of 50 mL SIG-001 spheres [an encapsulated allogeneic cell therapy genetically modified with a non-viral vector to produce B-Domain Deleted Human Factor VIII (BDD-hFVIII) producing Spheres] administered laparoscopically into the peritoneal cavity.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 1 | 1
  United Kingdom | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Number of Participants with at least one TEAEs are reported. A summary of other nonserious adverse events (AEs), and all serious adverse events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Up to 115 Weeks
Population: All participants who received at least one dose of study drug and have at least one postdose safety assessment.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 1
Participants | 1 | 1 | 1

2. Primary Outcome: Number of Participants With Serious Treatment Emergent Adverse Events (TEAEs)
Description: Number of Participants with at least one serious TEAEs are reported. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline Up to 115 Weeks
Population: All participants who received at least one dose of study drug and have at least one postdose safety assessment.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 1
participants | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Inhibitor Titer Values Assessed by Nijmegen Bethesda Assay
Description: Development of FVIII inhibitors is measured using the Nijmegen Bethesda inhibitor assay. The assay measures inhibitors to BDD-FVIII and also other forms of FVIII in the plasma, although rFVIII-BDD was used as a calibrator.
Time Frame: Baseline Up to 115 Weeks
Population: All participants who received at least one dose of study drug and had at least one postbaseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 1
participants | 0 | 0 | 1

4. Secondary Outcome: Change From Baseline in FVIII Activity Levels Assessed by One-stage and Chromogenic Assays
Description: The change from baseline in FVIII activity, as measured by one-stage and chromogenic assays) is summarized.
Time Frame: Baseline Up to 115 Weeks
Population: All participants who received at least one dose of study drug and had at least one postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: International Unit/deciliter (IU/dL)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 1
International Unit/deciliter (IU/dL)
  Chromogenic Assay | 13.03 (NA) — The number of participants is 1, so the Standard Deviation was not calculated. | 223.78 (NA) — The number of participants is 1, so the Standard Deviation was not calculated. | -122.71 (NA) — The number of participants is 1, so the Standard Deviation was not calculated.
  One-stage | 15.46 (NA) — The number of participants is 1, so the Standard Deviation was not calculated. | 118.28 (NA) — The number of participants is 1, so the Standard Deviation was not calculated. | 189.63 (NA) — The number of participants is 1, so the Standard Deviation was not calculated.

5. Secondary Outcome: Number of Bleeding Events [Annualized Bleeding Rate (ABR)] for All Bleeds Following SIG-001 Administration
Description: The annualized number of bleeds per participant (annualized bleeding rate) is calculated as the number of bleeding events divided by length of time on study product follow-up, in years. The duration of assessment for this outcome measure was two years and three months, and Year 3 includes only the three-month part of this study period.
Time Frame: Time Frame: Pre-infusion (bleeding events in 12 months prior to sphere placement), 1 year, 2 year and 3-year post-infusion (post sphere placement) from SIG-001 administration annualized up to 115 Weeks.
Population: All participants who received at least one dose of study drug and had at least one postbaseline efficacy assessment.
Measure: Number; unit: Bleeding events per year
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 1
Bleeding events per year
  Pre-infusion | 4 | 0 | 4
  Year 1 | 7 | 1 | 10
  Year 2 | 5 | 0 | 0
  Year 3 | 0 | 0 | NA — Data not available as participant left the study before year 3

6. Secondary Outcome: Total Number of Replacement FVIII Therapies
Description: Number of doses after prophylaxis discontinued is reported.
Time Frame: Baseline Up to 115 weeks
Population: All participants who received at least one dose of study drug and had at least one postbaseline efficacy assessment.
Measure: Number; unit: Number of doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 1
Number of doses | 401 | 327 | 1558

ADVERSE EVENTS:
Time Frame: Baseline Up to 115 Weeks
Description: All participants who received at least one dose of study drug.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=1) | Cohort 2 (N=1) | Cohort 3 (N=1)
Factor viii inhibition (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug ineffective (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anti factor viii antibody increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=1) | Cohort 2 (N=1) | Cohort 3 (N=1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cullen's sign (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT04541628/Prot_000.pdf